CLINICAL TRIAL: NCT04470102
Title: A Randomised Controlled Pilot Trial: Edge-to-edge Mitral Valve Repair in the Surgical Treatment for Hypertrophic Cardiomyopathy
Brief Title: Edge-to-edge Mitral Valve Repair in the Surgical Treatment for Hypertrophic Cardiomyopathy
Acronym: PRIZMA-pilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 188
Record Dates: First submitted 2020-07-08; First posted 2020-07-14 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: edge-to-edge repair; mitral valve plastic (MVP); Septal myectomy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial comparing mitral valve repair using the edge-to-edge technique for surgical treatment of hypertrophic cardiomyopathy
Masking Description: no data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isolated septal myectomy (Other): Isolated extended septal myectomy
  Interventions: Procedure: Septal myectomy
- Septal myectomy+ "edge-to-edge" (Active Comparator): advanced septal myectomy in combination with mitral valve repair using the edge-to-edge technique
  Interventions: Procedure: mitral valve repair by edge-to-edge technique

INTERVENTIONS:
Procedure: mitral valve repair by edge-to-edge technique — transaortic access for mitral valve repair edge-to-edge
  Other Names: Alfieri stitch
  Arms: Septal myectomy+ "edge-to-edge"
Procedure: Septal myectomy — isolated extended septal myectomy
  Other Names: Septal myectomy (SM)
  Arms: isolated septal myectomy

SUMMARY:
Objective of the study: to evaluate whether edge-to-edge technique improves clinical and hemodynamic results in patients scheduled to septal myectomy for severely symptomatic hypertrophic obstructive cardiomyopathy.

DETAILED DESCRIPTION:
A randomised controlled pilot trial to evaluate whether edge-to-edge technique improves clinical and hemodynamic results in patients scheduled to septal myectomy for severely symptomatic hypertrophic obstructive cardiomyopathy. Patients with proven hypertrophic cardiomyopathy and resting left ventricle outflow tract obstruction underwent septal myectomy. If patients were suitable for both surgical techniques, they were randomized to septal myectomy + edge-to-edge mitral valve repair or isolated septal myectomy. All surgeons were experienced at least 50 related procedures.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent (either from the patient or a substitute decision-maker)
* Indications for surgical treatment (septal myectomy) of hypertrophic cardiomyopathy

Exclusion Criteria:

* indications for mitral valve replacement
* Patient failure at any stage of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Outflow Tract (LVOT) gradient | 12 months in the medium-term follow-up
  Gradient at the level of the output section of the left ventricle after surgery (mmHg) This measurement will be performed by transthoracic echocardiography at rest and / or during exercise. The Doppler method will be used.

SECONDARY OUTCOMES:
Systolic anterior motion of the mitral valve | 12 months in the medium-term follow-up
  Systolic anterior motion of the mitral valve after surgery This measurement will be performed by transthoracic echocardiography at rest and / or during exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V. Bogachev-Prokophiev, MD, PhD, Principal Investigator — E.Meshalkin National medical research center
Locations (1):
- "E.Meshalkin National medical research center" of the Ministry of Health of the Russian Federation, Novosibirsk, Russia